CLINICAL TRIAL: NCT06397040
Title: The Use of Remote Monitoring to Improve Patient-Reported Outcomes and Readmission Rates Following Radical Cystectomy
Acronym: WATCH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Bruce Jacobs, Associate Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY23110094
Record Dates: First submitted 2024-04-23; First posted 2024-05-02 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-03

CONDITIONS: Bladder Cancer; Quality of Life
Keywords: bladder cancer; remote monitoring; quality of life; cystectomy
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- remote monitoring without provider feedback (Experimental): remote monitoring with FitBit device and daily patient-reported outcome assessment, without real-time provider feedback
  Interventions: Device: participant monitoring of remote data
- remote monitoring with provider feedback (Experimental): remote monitoring with FitBit device and daily patient-reported outcome assessment, as well as real-time provider feedback in response to remote data
  Interventions: Device: provider monitoring and feedback to remote data; Device: participant monitoring of remote data

INTERVENTIONS:
Device: provider monitoring and feedback to remote data — provider monitoring of remote data and feedback to changes in remote data
  Arms: remote monitoring with provider feedback
Device: participant monitoring of remote data — participant monitoring of remote data, based upon post-operative instructions

SUMMARY:
Following radical cystectomy for bladder cancer, nearly two-thirds of patients experience a complication and almost a third are readmitted. Thus, intensified monitoring of this vulnerable group represents an opportunity for improved quality of care in the post-operative setting. By gathering biomarkers passively and continuously, wearable activity monitors augment remote patient monitoring. Further, they facilitate the collection of patient-reported outcomes frequently.

Despite the proven impact of remote monitoring on patient care, there is limited data on the feasibility and impact of employing this technology to trigger real-time provider assessment following cystectomy. The investigators plan to conduct a randomized control trial examining such. The intervention group of participants will receive continuous biomarker monitoring via FitBits and daily patient-reported outcome assessments via connected smartphones. Abnormalities in remote data will trigger automated alerts to providers. Providers will respond in real-time to these alerts and patients will receive education materials discussing preventative measures to mitigate the main risk factors for readmissions. The investigators will evaluate the feasibility of integrating this technology into the post-operative period, as well as the impact of real-time provider attention to abnormal remote data on patient-reported outcomes and rates of readmission. The investigators hypothesize that early assessment of and intervention on remote abnormalities will promote the use of outpatient or reduced intensity therapies, such as oral antibiotics or oral hydration, thus curtailing the severity of patient symptoms, intensity of complications, and need for hospitalizations. Ultimately, this trial builds upon prior research, applying patient-centered technology to improve the quality of care following cystectomy.

ELIGIBILITY:
Inclusion Criteria:

* undergoing cystectomy at three hospitals within the University of Pittsburgh Medical Center system
* English speaking
* owns smart phone

Exclusion Criteria:

* unwilling or unable to participate
* non-English speaking
* does not own smart phone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
patient engagement | 4 weeks following hospital discharge
  percent of patients who utilized the application daily and wore the device for 8hrs daily
provider response | 4 weeks following hospital discharge
  time from alert to provider response to patient

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Marchetti, MD, Principal Investigator — University of Pittsburgh Medical Center
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The data will be available at the time of publication and 7 years following (as data stored at institution for 7 years following project completion.
Access Criteria: Interested researcher can contact the study team for individual participant data. The data will be made available following data use agreement.